CLINICAL TRIAL: NCT04056091
Title: Back Rubs or Foot Flicks for Neonatal Stimulation at Birth in a Low-resource Setting: an Open-label Randomised Superiority Trial
Brief Title: Back Rubs or Foot Flicks for Neonatal Stimulation at Birth in a Low-resource Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Padova (Other)
Collaborators: Jerry Ictho (Unknown); John Bosco Nsubuga (Unknown); Jesca Ameo (Unknown); Giovanni Putoto (Unknown); Peter Lochoro (Unknown)
Responsible Party: Principal Investigator, Daniele Trevisanuto, Professor, University of Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRRH-REC OUT0017/2019
Record Dates: First submitted 2019-08-07; First posted 2019-08-14 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Neonatal Resuscitation
Keywords: Neonatal resuscitation; Stimulation; Asphyxia
MeSH Terms: conditions — Asphyxia

STUDY DESIGN:
Masking Description: Only statistician will be masked to tretament
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Back rub stimulation (Experimental)
  Interventions: Procedure: Back rub stimulation
- Foot flicks stimulation (Active Comparator)
  Interventions: Procedure: Foot flicks stimulation

INTERVENTIONS:
Procedure: Back rub stimulation — Immediately after birth, all infants with an expected birthweight >1500 g who have been dried and remain apneic (not crying) will receive physical stimulation (back rubs). Stimulation can be repeated at maximum two or three times for about 3-5 seconds.
  Arms: Back rub stimulation
Procedure: Foot flicks stimulation — Immediately after birth, all infants with an expected birthweight >1500 g who have been dried and remain apneic (not crying) will receive physical stimulation (foot flicks). Stimulation can be repeated at maximum two or three times for about 3-5 seconds.
  Arms: Foot flicks stimulation

SUMMARY:
Physical stimulation is the most common intervention during neonatal stabilization/resuscitation at birth and is recommended by neonatal resuscitation guidelines in high as well low-income settings. Two modalities of stimulation (back rubs or foot flicks) are recommended.

This is a single center, unblinded, randomized superiority trial. Immediately after birth, all "not crying" infants will be randomly assigned in a 1:1 ratio to two different modes of stimulation (back rubs or foot flicks). Exclusion criteria will be stillbirths and presence of major neonatal malformations. The primary outcome measure will be the need for FMV. Secondary outcome measures will include Apgar score at 5 minutes, time of initiation and duration of FMV, time to first cry (defined as the first audible cry spontaneously emitted by the infant), death or moderate to severe hypoxic-ischemic encephalopathy within 7 days of life or at discharge, admission to special care, and procedure-associated complications.

The results of the present study will help to identify the most appropriate mode for stimulating the apneic newly infants in delivery room. In clinical practice, this information is very relevant because effective stimulation at birth will elicit spontaneous respiratory in a certain percentage of apneic neonates avoiding the need for positive pressure ventilation and, possibly, further advanced resuscitative maneuvers.

ELIGIBILITY:
Inclusion Criteria:

1. Newly born infants who are apneic (not crying) immediately after birth (and)
2. Expected birthweight > 1500 g (and)
3. Parental consent

Exclusion Criteria:

1. Still births
2. Twins
3. Major congenital malformations (i.e. congenital cardiac malformation, pulmonary hypoplasia, major spina bifida, etc.)

Ages: 1 Minute to 10 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 186 (Estimated)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of babies needing positive pressure ventilation | 2 minutes

SECONDARY OUTCOMES:
Apgar score at 5 minutes | 5 minutes
  Apgar score is a scale from 0 (very bad) to 10 (very good) that classify the clinical condition of the neonates during the first minutes of life
Time of initiation of face-mask ventilation | 5 minutes
Time of duration of face-mask ventilation | 20 minutes
Time to first cry | 20 minutes
Percentage of deaths | 7 days
Peercentage of babies admitted to special care | 2 hours
Percentage of procedure-associated complications | 3 days
Percentage of babies with moderate to severe hypoxic-ischemic encephalopathy | 7 days
  The grade of encephalopathy will be measured according to a modified Sarnat and Sarnat classification

CONTACTS AND LOCATIONS:
Locations (1):
- Matany Hospital, Moroto, Karamoja, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dekker J, Martherus T, Cramer SJE, van Zanten HA, Hooper SB, Te Pas AB. Tactile Stimulation to Stimulate Spontaneous Breathing during Stabilization of Preterm Infants at Birth: A Retrospective Analysis. Front Pediatr. 2017 Apr 3;5:61. doi: 10.3389/fped.2017.00061. eCollection 2017. PMID 28421171
- [Result] Owen CJ, Wyllie JP. Determination of heart rate in the baby at birth. Resuscitation. 2004 Feb;60(2):213-7. doi: 10.1016/j.resuscitation.2003.10.002. PMID 15036740
- [Result] Voogdt KG, Morrison AC, Wood FE, van Elburg RM, Wyllie JP. A randomised, simulated study assessing auscultation of heart rate at birth. Resuscitation. 2010 Aug;81(8):1000-3. doi: 10.1016/j.resuscitation.2010.03.021. Epub 2010 May 18. PMID 20483522
- [Result] Pietravalle A, Cavallin F, Opocher A, Madella S, Cavicchiolo ME, Pizzol D, Putoto G, Trevisanuto D. Neonatal tactile stimulation at birth in a low-resource setting. BMC Pediatr. 2018 Sep 20;18(1):306. doi: 10.1186/s12887-018-1279-4. PMID 30236090
- [Result] Gaertner VD, Flemmer SA, Lorenz L, Davis PG, Kamlin COF. Physical stimulation of newborn infants in the delivery room. Arch Dis Child Fetal Neonatal Ed. 2018 Mar;103(2):F132-F136. doi: 10.1136/archdischild-2016-312311. Epub 2017 Jun 9. PMID 28600392
- [Result] Wyllie J, Bruinenberg J, Roehr CC, Rudiger M, Trevisanuto D, Urlesberger B. European Resuscitation Council Guidelines for Resuscitation 2015: Section 7. Resuscitation and support of transition of babies at birth. Resuscitation. 2015 Oct;95:249-63. doi: 10.1016/j.resuscitation.2015.07.029. Epub 2015 Oct 15. No abstract available. PMID 26477415
- [Result] Kamath-Rayne BD, Berkelhamer SK, Kc A, Ersdal HL, Niermeyer S. Neonatal resuscitation in global health settings: an examination of the past to prepare for the future. Pediatr Res. 2017 Aug;82(2):194-200. doi: 10.1038/pr.2017.48. Epub 2017 May 24. PMID 28419084
- [Result] Wyckoff MH, Aziz K, Escobedo MB, Kapadia VS, Kattwinkel J, Perlman JM, Simon WM, Weiner GM, Zaichkin JG. Part 13: Neonatal Resuscitation: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S543-60. doi: 10.1161/CIR.0000000000000267. No abstract available. PMID 26473001
- [Derived] Cavallin F, Lochoro P, Ictho J, Nsubuga JB, Ameo J, Putoto G, Trevisanuto D. Back rubs or foot flicks for neonatal stimulation at birth in a low-resource setting: A randomized controlled trial. Resuscitation. 2021 Oct;167:137-143. doi: 10.1016/j.resuscitation.2021.08.028. Epub 2021 Aug 23. PMID 34438002
- See also: Related Info — http://www.helpingbabiesbreathe.org
- See also: Related Info — http://www.cuamm.org